CLINICAL TRIAL: NCT06906549
Title: Evaluation of 200 mg of Rituximab Every 6 Months as Maintenance Treatment of Rituximab-treated Patients With Rheumatoid Arthritis: a Non-inferiority Prospective Randomised Controlled Trial
Brief Title: Evaluation of 200 mg of Rituximab Every 6 Months as Maintenance Treatment of Rituximab-treated Patients With Rheumatoid Arthritis
Acronym: RADAR
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 9424; 2024-519991-18-00 (EU CTIS Number)
Record Dates: First submitted 2025-03-18; First posted 2025-04-02 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Rheumatoid Arthritis (RA); Rituximab (RTx)
Keywords: Dose reduction; Low dose Rituximab
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Rituximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rituximab 200mg/6months (Experimental)
  Interventions: Drug: Rituximab 200mg/6months
- Rituximab 1g/6 months (Active Comparator)
  Interventions: Drug: Rituximab 1g/6months

INTERVENTIONS:
Drug: Rituximab 200mg/6months — perfusion of Rituximab 200mg
  Arms: Rituximab 200mg/6months
Drug: Rituximab 1g/6months — perfusion of Rituximab 1g
  Arms: Rituximab 1g/6 months

SUMMARY:
Rheumatoid arthritis (RA) is a chronic inflammatory disease affecting joints and causing progressive disability. Current treatment strategies involve conventional disease-modifying anti-rheumatic drugs (csDMARDs) and, in more resistant cases, biologic DMARDs (bDMARDs) such as Rituximab. Rituximab, a monoclonal antibody targeting CD20-positive B cells, is administered as an induction dose followed by maintenance therapy every six months. Standard maintenance dosing consists of 1g infusions, but lower doses may provide equivalent efficacy with fewer side effects.

The RADAR trial is a multicenter, prospective, randomized, double-blinded, non-inferiority controlled trial designed to evaluate whether a 200 mg maintenance dose of Rituximab every six months is non-inferior to the standard 1g dose in patients with RA who are in low disease activity. The study will assess disease activity using the DAS28-CRP score over 12 months, alongside various secondary endpoints, including treatment failure rates, immune responses, and adverse events.

By determining the minimum effective Rituximab dose, the study aims to optimize patient safety, reduce the risk of infections, and lower healthcare costs. This trial is particularly relevant as Rituximab has lost patent protection, making cost-effective treatment crucial, especially in low-resource settings. Findings from this study could lead to updated treatment guidelines, benefiting RA patients worldwide.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is the most prevalent chronic inflammatory rheumatic disease in Europe, affecting 0.3%-0.5% of the population. Treatment follows a Treat-to-Target (T2T) approach, where patients are initially managed with conventional synthetic DMARDs (csDMARDs), such as methotrexate, and if necessary, escalated to biologic DMARDs (bDMARDs) like Rituximab, a monoclonal antibody that depletes CD20-positive B cells.

The current standard maintenance therapy for RA patients receiving Rituximab consists of 1g infusions every six months. However, concerns about long-term safety, immune suppression, and cost have led researchers to explore lower doses. Studies suggest that 200 mg of Rituximab may be sufficient to maintain disease control while potentially reducing the risks associated with B-cell depletion, such as hypogammaglobulinemia and serious infections.

Study Rationale and Objectives The RADAR trial aims to provide definitive evidence on the feasibility of reducing Rituximab doses without compromising efficacy. A previous randomized trial indicated that a 500 mg dose was non-inferior to 1g, but the 200 mg arm lacked sufficient statistical power. Subsequent long-term follow-up data suggest that 200 mg may also be effective, warranting further investigation.

The primary objective of this study is to demonstrate that the 200 mg Rituximab maintenance dose is non-inferior to 1g in terms of disease activity, measured by DAS28-CRP at 12 months.

Secondary objectives include:

* Comparing disease activity at 6 and 12 months
* Evaluating treatment failure rates (need for additional Rituximab doses, switching to other bDMARDs, corticosteroid use)
* Assessing flare occurrence and patient-reported outcomes (quality of life, disability index)
* Investigating B and T lymphocyte subpopulations and immunoglobulin levels (IgG, IgA, IgM)
* Analyzing vaccine responses and Human Anti-Chimeric Antibody (HACA) levels
* Monitoring immunosuppression markers, such as Torque Teno Virus (TTV) viral load
* Documenting adverse and serious adverse events Study Design

This is a multicenter, double-blinded, non-inferiority, randomized controlled trial (RCT). Patients will be randomized 1:1 to receive either:

1. 200 mg of Rituximab (experimental group)
2. 1g of Rituximab (control group) Participants will receive two infusions: one at baseline (Month 0) and one at 6 months, with follow-up visits at 4, 6, 10, and 12 months. The primary endpoint is the mean reduction in DAS28-CRP between baseline and 12 months.

Blinding Procedure:

* Infusions will be prepared in the central pharmacy to ensure identical appearance in both groups.
* Neither patients nor clinicians will know the assigned dosage.

Inclusion criteria:

* Adults (≥18 years) with RA (EULAR/ACR 2010 criteria)
* Low disease activity (DAS28-CRP <3.2) on Rituximab
* Prior treatment with Rituximab (at least one infusion in the past year)
* Stable on csDMARDs (if applicable)
* Corticosteroid dose ≤10 mg/day

Non-inclusion criteria:

* Autoimmune diseases other than RA
* Severe infections, immunodeficiency, or uncontrolled disease
* Active or untreated tuberculosis, hepatitis B/C
* Pregnancy, breastfeeding, or planned pregnancy
* Drug/alcohol addiction
* Patients unable to give informed consent Study Assessments and Data Collection

The study will include clinical, biological, and immunological assessments:

* DAS28-CRP scores at baseline, 6, and 12 months
* Immunological assays (B/T cell phenotyping, immunoglobulin levels, HACA)
* Vaccine serologies (Diphtheria, Pneumococcus, Tetanus, Haemophilus, SARS-CoV-2)
* Quality-of-life surveys (EQ-5D-5L, SF-36, RAPID-3)
* Adverse event monitoring

Sample Size Calculation:

The trial requires 260 patients to achieve 92% power to detect non-inferiority, using a linear mixed model with a non-inferiority margin of -0.3 on DAS28-CRP.

Expected Impact

If 200 mg of Rituximab proves non-inferior to 1g, this study could redefine maintenance therapy guidelines, reducing:

* Drug exposure and immune suppression risks
* Serious infections and adverse events
* Healthcare costs, improving access in resource-limited settings By providing definitive clinical and immunological data, the RADAR trial has the potential to influence global RA management and enhance long-term treatment safety.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of rheumatoid arthritis (RA) according to EULAR/ACR 2010 classification criteria
* DAS28 ≤ 5.1
* Current maintenance treatment with Rituximab regardless of dose and/or duration of Rituximab treatment and with at least first cycle of Rituximab ended (2 initial infusions)
* Last Rituximab infusion between 6 and 18 months prior to inclusion
* Corticosteroids ≤10 mg/day within 4 weeks prior to inclusion
* Affiliation to a social insurance system or beneficiary
* Written informed consent to participate in the study, dated and signed before starting the trial
* Effective method of birth control during the study

Exclusion Criteria:

* Rheumatic autoimmune disease other than RA (except associated Sjogren's disease, which is allowed)
* Concurrent treatment with any other targeted therapy than Rituximab
* Any contraindication to Rituximab or to NaCl 0.9%
* Significant uncontrolled associated disease or comorbidity
* Known active infection or history of serious recurrent or chronic infection
* Laboratory findings: active or untreated latent tuberculosis, hepatitis B positive, hepatitis C positive, haemoglobin <8 g/dL, neutropenia < 1.5G/L, IgM <0.4 g/L and/or IgG <5 g/L
* Pregnancy, breastfeeding, or planned pregnancy during the study (on subject declaration)
* Drug addiction, alcohol addiction
* Patients who cannot be followed for the 12 month-duration
* Patients over the age of legal majority who are protected, or deprived of liberty by judicial or administrative decision
* Subject in exclusion period (determined by a previous or ongoing study)
* Patients unable to give informed consent (e.g., patients in a situation of medical emergency, patients who have difficulty comprehending the essential details of the trial...)
* Patients who have difficulty reading or understanding French, or who have an inability to understand the delivered information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2025-07-11 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Mean reduction of rheumatoid arthritis activity score (DAS28-CRP) | 12 Months
  Mean reduction of rheumatoid arthritis activity score (DAS28-CRP) between inclusion and 12 months to show non-inferiority of the lower dose.

SECONDARY OUTCOMES:
Compare the disease activity measured by DAS28-CRP between the two arms | at inclusion, 6 and 12 months
DAS28 categories | at inclusion, 6 months and 12 months
  Remission: DAS28 < 2.6 ; Low Disease Activity: 2.6 ≤ DAS28 ≤ 3.2 ; Moderate Activity: 3.2 < DAS28 ≤ 5.1; High Disease Activity: DAS28 > 5.1 ; Boolean Remission Criteria defined as tender joint count (TJC) ≤ 1, swollen joint count (SJC) ≤ 1, CRP (mg/dL) ≤ 1, Patient global assessment (on a 0-10 scale) ≤ 1
Number of Rituximab infusions | 12 Months
Number of patients switching or initiating a cDMARD or switching from Rituximab to another bDMARD | 12 Months
Number of patients using oral corticosteroids at a dose greater than 10 mg/day | 12 Months
Number of flares throughout study period | 12 Months
FLARE questionnaire (FLARE ASSESSMENT IN RHEUMATOID ARTHRITIS) | at 6 and 12 months
  FLARE-RA is a self-administered questionnaire that was developed to help identify patients who had flare in the interval between 2 rheumatology consultations. To establish a threshold for the FLARE-RA score to identify RA flare.
RAPID-3 score (ROUTINE ASSESSMENT OF PATIENT INDEX DATA 3) | at inclusion, 6 and 12 months
  RAPID3 : Index to asses and monitor patients with RA
RAID score (RHEUMATOID ARTHRITIS IMPACT OF DISEASE) | at inclusion, 6 and 12 months
  The Rheumatoid Arthritis Impact of Disease (RAID) score is a EULAR-initiated PROM developed in collaboration with patients with RA. It is a global composite measure of the impact of RA that takes into account: pain, physical disability, fatigue, sleep disturbances, coping as well as physical and emotional well-being.
  The RAID score was calculated using the online EULAR toolkit. Each of the seven individual domains of the RAID is scored on a 10-item numerical rating scale, with zero being a good or low activity score and 10 a high or severe activity score. In the absence of guidance, we arbitrarily classified the numerical rating scale results into one of three equivalent-sized ranges (mild: 0-2; moderate: 3-6; severe: 7-10) to give an overall idea of which domains scored particularly poorly or well.
EQ5D-5L (EUROQOL GROUP) | at inclusion, 6 and 12 months
  The EQ-5D family of instruments has been developed to describe and value health across a wide range of disease areas. They are frequently used in research into health in the general population. There are three versions of the instrument: EQ-5D-5L, EQ-5D-3L and EQ-5D-Y. The EQ-5D is used worldwide and has been translated into most major languages through a closely monitored translation process.
  The 5-level EQ-5D version (EQ-5D-5L) consists of 2 tests: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).
  * The EQ-5D-5L descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression.
  * The EQ VAS records the patient's self-rated health on a vertical visual analogue scale where the endpoints are labelled 'Best imaginable health state' =100 and 'Worst imaginable health state'=0.
SF-36 to compare the patient quality of life | at inclusion, 6 and 12 months
  SF-36 (MEDICAL OUTCOMES STUDY SHORT FORM HEALTH SURVEY 36 - RAND CORPORATION)
B, T and NK cell phenotyping to compare cell subpopulations | at inclusion, 6 and 12 months
Compare change in IgG, IgA and IgM levels | at inclusion, 6 and 12 months
Vaccinal serologies to compare vaccine response | at inclusion, 6 and 12 months
  Diphteria, pneumococcus, tetanus, Haemophilus influenzae type B and SARS-CoV-2
Compare HACA (Human antichimeric antibody) levels | at inclusion and 12 months
Evolution of Torque Teno Virus (TTV) viral load in the serum of patients | between inclusion and 12 months
Number of infections | 12 Months
Number of serious infections | 12 Months
Number of adverse events | 12 Months
Number ofserious adverse events | 12 Months

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpitaux Universitaires de Strasbourg, Strasbourg, France